CLINICAL TRIAL: NCT01446848
Title: Oral Iron Supplementation in Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Samar Farha, MD, Staff Pulmonologist, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPC-2011-1026
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: iron deficiency; pulmonary hypertension; iron supplements; ferrous sulfate
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Iron Deficiencies; Hypertension, Pulmonary | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iron supplement (Experimental): open-label iron supplement intervention group
  Interventions: Dietary Supplement: iron supplement

INTERVENTIONS:
Dietary Supplement: iron supplement — 325 mg tablets by mouth once a day for 1 week, then twice a day for 1 week, then three times daily for the remainder of the 3-month study period.
  Other Names: ferrous sulfate tablets

SUMMARY:
The purpose of this study is to investigate the effects of iron supplementation in patients with pulmonary arterial hypertension and iron deficiency.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a chronic disease associated with upregulation of hypoxia inducible-factor-1alpha (HIF-1alpha) and functional iron deficiency. The investigators are proposing a prospective, single-arm, open-label intervention to determine whether oral iron supplementation in patients with pulmonary arterial hypertension reduces markers of HIF activation and improve clinical parameters of disease. After the baseline visit, patients will be given ferrous sulfate tablets to take orally for 3 months. Outcome data will be collected at the baseline visit and at the end of the 3-month study period.

ELIGIBILITY:
Inclusion Criteria:

* age 21 and older
* diagnosis of idiopathic pulmonary arterial hypertension
* iron deficiency (transferrin saturation <20% and serum ferritin < 100 ug/l)

Exclusion Criteria:

* active infection, malignancy, or bleeding
* hemochromatosis
* chronic inflammatory or autoimmune disease
* currently taking experimental/study medications, erythropoietin, iron supplementation, or immunosuppressants
* allergy to iron

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in Zinc protoporphyrin from baseline | 3 months
Change in serum ferritin from baseline | 3 months

SECONDARY OUTCOMES:
Change in serum erythropoietin from baseline | 3 months
Change in transferrin saturation from baseline | 3 months
Change in %CD34+/133+ cells from baseline | 3 months
Change in pulmonary arterial pressure from baseline | 3 months
  estimated using echocardiogram
Change in six minute walk distance from baseline | 3 months
NYHA/WHO classification | 3 months
Side effects of iron supplementation | 3 months
Deaths and hospitalizations greater than 24 hours | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Samar Farha, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States